CLINICAL TRIAL: NCT04890730
Title: Southern Medical University of Nanfang Hospital
Brief Title: Non-invasive Method for Predicting the Presence of Gastroesophageal Varices in Patients With Cirrhosis-a Prospective, Multicenter Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2020-222
Record Dates: First submitted 2021-05-10; First posted 2021-05-18 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Gastroesophageal Varices; Decompensation Event
MeSH Terms: interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Take 10ml blood sample for each patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Southern Medical University of Nanfang Hospital: Southern Medical University of Nanfang Hospital
  Interventions: Other: Esophagogastroduodenoscopies
- Tongji Hospital Affiliated to Tongji University: Tongji Hospital Affiliated to Tongji University
  Interventions: Other: Esophagogastroduodenoscopies
- The Second Affiliated Hospital Of Nanchang University: The Second Affiliated Hospital Of Nanchang University
  Interventions: Other: Esophagogastroduodenoscopies

INTERVENTIONS:
Other: Esophagogastroduodenoscopies — Each enrolled patient needs to undergo Esophagogastroduodenoscopies and elastography

SUMMARY:
Gastroesophageal varices are a complication of portal hypertension in cirrhosis.Endoscopy is an unsatisfactory screening test.In this prospective clinical study,we will enroll patients with cirrhosis of various causes, all of whom undergo laboratory tests, elastography, and serum proteomic differential protein testing, including liver elastography (LSM) and spleen elastography (SSM). Baveno VI or expanded BavenoVI criteria are validated by comparing patients' LSM and PLT. LSM, SSM, serum differential protein, platelet count, and EGD data to evaluate the clinical value of SSM and differential proteins in excluding cirrhosis with varices. At the same time, a new predictive model of variceal varices will be established to evaluate the diagnostic value of SSM and differential protein for esophagogastric varices, and a non-invasive method for reliably predicting and evaluating cirrhosis with esophageal varices will be found. And each patient will be followed up every 6 months to 1 year, and the outcome event will be recorded.

DETAILED DESCRIPTION:
Gastroesophageal varices are a complication of portal hypertension in cirrhosis.Endoscopy is invasive method as an unsatisfactory screening test.In this prospective clinical study, we will enroll patients with cirrhosis of various causes, all of patients whom undergo laboratory tests, elastography, and serum proteomic differential protein testing, including LSM and SSM. Baveno VI or expanded BavenoVI criteria are validated by comparing patients' LSM and PLT. LSM,SSM, serum differential protein, platelet count, and EGD data to evaluate the clinical value of SSM and differential proteins in excluding cirrhosis with varices. At the same time, based on SSM and serum differential protein, a new predictive model of variceal varices will be established to evaluate the diagnostic value of SSM and differential protein for esophagogastric varices, and a non-invasive method for reliably predicting and evaluating cirrhosis with esophageal varices will be found. And each patient will be followed up every 6 months to 1 year, and the outcome event will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 1. The age ranged from 18 to 80 years. 2. Clinical or pathological diagnosis of cirrhosis; 3. Electronic gastroscopy is planned; 4. To agree and sign the informed consent;

Exclusion Criteria:

* 1.Orthotopic liver transplantation patients; 2. Patients who have undergone transjugular intrahepatic portosystemic shunt (TIPS),or previous surgical shunt; 3. Pregnant women; 4. Neurological or psychiatric disorders;

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who come to the center to see a doctor who meet the enrollment criteria and agree to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 992 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of high-risk esophageal varices | 4 years
  Incidence of high-risk esophageal varices

SECONDARY OUTCOMES:
Incidence of hemorrhagic events | 4 years
  Incidence of hemorrhagic events
Incidence of Clinical decompensation events and deaths | 4 years
  Incidence of Clinical decompensation events and deaths

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatology Unit, Department of Infectious Diseases, Nanfang Hospital, Southern Medical University, Guangzhou, China

REFERENCES:
- [Derived] Zhang X, Song J, Zhang Y, Wen B, Dai L, Xi R, Wu Q, Li Y, Luo X, Lan X, He Q, Luo W, Lai Q, Ji Y, Zhou L, Qi T, Liu M, Zhou F, Wen W, Li H, Liu Z, Chen Y, Zhu Y, Li J, Huang J, Cheng X, Tu M, Hou J, Wang H, Chen J. Baveno VII algorithm outperformed other models in ruling out high-risk varices in individuals with HBV-related cirrhosis. J Hepatol. 2023 Mar;78(3):574-583. doi: 10.1016/j.jhep.2022.10.030. Epub 2022 Nov 7. PMID 36356684